CLINICAL TRIAL: NCT00959816
Title: A Study to Investigate the Process by Which ABT-614 is Absorbed, Distributed, Metabolized and Eliminated in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Beatrice Rendenbach-Mueller, PhD / Project Director, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M11-954
Record Dates: First submitted 2009-08-13; First posted 2009-08-17 (Estimated); Last update posted 2010-11-02 (Estimated); Status verified 2010-09

CONDITIONS: Healthy
Keywords: Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single Dose (Part 1) (Experimental)
  Interventions: Drug: ABT-614
- Multiple Dose (Part 2) (Experimental)
  Interventions: Drug: ABT-614

INTERVENTIONS:
Drug: ABT-614 — Single dose administered on Study Day 1 in Part 1, daily dose administered on Study Days 1-14 in Part 2.

SUMMARY:
The objective of this study is to determine the amount of ABT-614 in the cerebral spinal fluid and blood after administration of a single dose and after administration of daily doses for 14 days in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between 18 and 40 years of age

Exclusion Criteria:

* History of bleeding disorders or deep vein thrombosis (DVT)
* Previous gastrointestinal (GI) surgery or chronic GI disease
* History of spinal surgery
* History of significant, chronic low back pain
* History of frequent headaches

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2009-08; Primary Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability Assessments (e.g., clinical laboratory tests, vital signs, adverse event assessment, physical examination) | One day before dosing through day of last dose and up to 72 hrs post-single dose or up to 14 days post-multiple doses
ABT-614 levels in cerebral spinal fluid | 0-24 hrs after single dose or 0-24 hrs after last dose of mulitple-dosing regimen
ABT-614 levels in blood (plasma) | 0-24 hrs after single dose or 0-24 hrs after last dose of mulitple-dosing regimen

CONTACTS AND LOCATIONS:
Locations (1):
- Site Reference ID/Investigator# 22445, San Antonio, Texas, United States